CLINICAL TRIAL: NCT01886560
Title: Prospective, Double-blind, Randomized, Controlled Clinical Trial of Low Dose Doxycycline in the Treatment of Corneal Burn
Brief Title: Low Dose Doxycycline in the Treatment of Corneal Burn
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dan Liang, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SunYat-senU2
Record Dates: First submitted 2013-06-14; First posted 2013-06-26 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-06

CONDITIONS: Eye Burns
MeSH Terms: conditions — Eye Burns | interventions — Doxycycline; sulfadiazine, tetroxoprim drug combination; Chlortetracycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Adding eatable flour into the pills
  Interventions: Drug: Placebo
- Doxycycline treatment (Experimental): Doxycycline treatment 50mg bid x 14 days then 50mg qd x 10 weeks
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — Tablets Doxycycline 50mg bid for 2 weeks,50mg qd for 10 weeks.
  Other Names: Dolotard; Tibirox; Biomycin
  Arms: Doxycycline treatment
Drug: Placebo — Tablets placebo one PO per day for 12 weeks
  Other Names: dummy
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of oral low dose doxycycline in the treatment of corneal burn.

DETAILED DESCRIPTION:
Severe Ocular Burn often leads to the Ocular surface failure, corneal vascularization dissolved hole or corneal opacity.Because the conventional treatment effect is not ideal, blindness rate is extremely high, has been a very challenging catastrophic ophthalmic emergency.Early effective inhibition of inflammation, promote healing of corneal epithelium is the key of reducing corneal perforation, corneal neovascularization, improving corneal transparency.Existing anti-inflammatory treatment including the hormone and immune inhibitors, auto-serum, non-steroidal anti-inflammatory drugs, amniotic membrane transplantation or amniotic membrane patch, etc.Although these measures have some effect, they have their disadvantages.Select both broad-spectrum anti-inflammatory effects and moderate price, good safety anti-inflammatory drugs is particularly important.

Sub-antimicrobial dose doxycycline posses known anti-inflammatory effects that are separate from their antibacterial mode of action.This mode of action has lead to the routine use of sub-antimicrobial dose doxycycline for treating inflammatory or autoimmune diseases, such as rosacea, periodontitis and multiple sclerosis.We confirmed on the basis of predecessors' studies that low dose oral doxycycline and topical application of doxycycline can accelerate corneal epithelium healing after ocular surface burn, effectively inhibit inflammation mediated corneal new angiogenesis.Its mechanism of action is about downregulate MMP2 and nitric oxide synthase.

Given the previous research obtained the encouraging result, we plan to carry out a clinical research, to explore oral low-dose doxycycline efficacy and safety of the treatment of corneal burns.

ELIGIBILITY:
Inclusion Criteria:

* 1.age from 18-70 years old, not limited to sex

  2. ocular burn (including chemical injury, thermal burns)

  3. studies of eye with Dua grade (2001) III, within 14 days after burns

  4. about the eye burns
  1. become the research with only one eye
  2. conform to the standards of subjects for the eyes

Choose poor eyesight as in the study

If the vision is the same on both sides, the choice classification is higher as the research of eye

If the binocular vision and graded at the same time, according to a study in can be determined in consultation with the patient's eye

5.signed informed consent form

Exclusion Criteria:

- 1. Only one eye function

2.The exclusion criteria of the eye

A) corneal thinning depth ≥ 1/2CT, corneal perforation or perforation tendency

B, Dua classification I、II、IV、V、VI

C) after injury had received eye operation (such as amniotic membrane transplantation or covering)

D) Poor control of intraocular pressure after anti-glaucoma drug treatment (IOP ≥ 25mmHg)

E) past other corneal diseases

F) past ocular history of radiation therapy or eye operation history

G) eyelid defect, incomplete eyelid closure, entropion, trichiasis

3. Any side formulated after secondary infection

4. Other rule out criteria

A) Tetracycline class history of drug allergy

B) poor control of blood pressure (defined as after treatment with antihypertensive drugs, blood pressure is 150/95mmHg or higher)

C) serious heart, hepatic, renal insufficiency (or myocardial infarction, arrhythmia, myocardial ischemia and cardiac insufficiency, ALT, AST, upper limit of normal or higher by 2.5 times, creatinine upper limit of normal or higher by 1.5 times)

D) during pregnancy or lactation women (defined as pregnancy urine pregnancy test results in this test)

E) child-bearing age subjects (male and female) is suitable precautions during the entire study

F) into the group participated in other clinical subjects before 3 months

G) people with TB

H) nerve with mental illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Time for Corneal epithelialization after treatment | 24 weeks

SECONDARY OUTCOMES:
corneal limbal ischemia | 12 weeks
Safety and tolerability as assessed by adverse events, vital signs | 24 weeks
corneal neovascularization | 12 weeks
Corneal transparency | 12 weeks
cornea ulcer with perforation | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dan Liang, MD, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, China
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China